CLINICAL TRIAL: NCT04990102
Title: Phase IB/II of CPX-351 as Maintenance Therapy in AML Patients Ineligible for Bone Marrow Transplantation
Brief Title: Phase IB/II of CPX-351 for Relapse Prevention in AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Jazz Pharmaceuticals (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003287
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia (AML) in Remission
Keywords: Acute Myeloid Leukemia; Remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351

STUDY DESIGN:
Intervention Model Description: Dose de-escalation of CPX-351
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-351 (Experimental): Dose Level 1: CPX-351 administered through intravenou infusion on Day 1 and Day 3 of 28 day cycle for 6 cycles or Dose Level -1: CPX-351 administered through intravenous infusion on Day 1 of each 28 day cycle for 6 cycles.
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — Daunorubicin 8.8mg/m2 + cytarabine 20mg/m2
  Other Names: Vyxeos

SUMMARY:
This is a phase IB/II study with a 3+3 dose de-escalation study design. Patients will continue maintenance treatment with CPX-351 for 6 cycles on D1 and D3, as long as patient remains in CR. The dose de-escalation will be one dose given on D1 only, every 28 days pending toxicity. The maximum tolerated dose will be used for the phase II expansion portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients > 18 years of age
* Patients must be in CR or CRh (complete remission with partial count recovery).
* Must have received ANY induction treatment with standard consolidation or hypomethylating agent (HMA) + venetoclax, for up to 6 cycles or no more than one year of treatment.
* Must be able to start therapy within 3 months of last documented CR
* De novo or secondary AML/treatment related AML (non-M3) including AML with myelodysplasia-related changes (MRC), histologically confirmed
* Patients must be ineligible for allogeneic BMT (for any reason including poor performance status, patient's preference, favorable AML not a candidate for transplant, or comorbidities and age precluding from transplant etc)
* Cardiac ejection fraction ≥ 50% by transthoracic echocardiography or MUGA scan
* Adequate hepatic and renal function defined as:

  * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 3 x upper limit of normal (ULN)
  * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 3 is permissible if due to disease.
  * Bilirubin ≤3 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
  * Estimated Creatinine Clearance ≥30 ml/min (Cockcroft-Gault based on actual weight) (See Appendix A)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 3 (Appendix A)
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry.
* Male and female subjects who agree to use highly effective methods of birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the period of therapy and for at least 6 months after the last dose of study drug

Exclusion Criteria:

* Prior allogeneic transplant
* Previous cumulative anthracycline (doxorubicin equivalent) dose equal to or greater than 345 mg/m2, and for patients with prior mediastinal XRT, anthracycline dose equal to or greater than 295 mg/m2
* Acute promyelocytic leukemia [t(15;17)]
* If patient is unable to sign informed consent due to any serious medical condition, laboratory abnormality or psychiatric illness
* Patients with evidence of uncontrolled current myocardial impairment (e.g. unstable ischemic heart disease, uncontrolled arrhythmia, symptomatic valvular dysfunction not controlled on medical therapy, uncontrolled hypertensive heart disease, and uncontrolled congestive heart failure)
* History of Wilson's disease or other copper-related disorders
* History of allergic reactions attributed to compounds of similar composition to cytarabine and daunorubicin or liposomal products
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4.03), grade ≤1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* Known active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, hepatitis C antibody, must have a negative polymerase chain reaction (PCR) result for the respective disease before enrollment. Those who are PCR positive will be excluded.
* Any uncontrolled active systemic infection.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* Known CNS involvement by leukemia
* Erythema multiforme, toxic epidermal necrolysis, or Stevens-Johnson syndrome
* Lactating or pregnant.
* Unwilling or unable to participate in all required study evaluations and procedures.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).
* Currently active, clinically significant hepatic impairment (≥ moderate hepatic impairment according to the Child Pugh classification (class B or C))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerate dose (Phase 1) | 1 cycle (28 day cycle)
  Number of subjects with Dose Limiting toxicities will be used to determine the recommended phase II dose of CPX-351 to be used in the maintenance setting for newly diagnosed AML in complete remission.
Inicidence of Treatment Emergent Adverse events (Phase 2) | 6 cycles (28 day cycles)
  To determine the safety, tolerability and toxicity of CPX-351 in the maintenance setting for newly diagnosed AML in complete remission by analyzing the incidence of treatment emergent adverse events reported.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (Phase 1) | 6 cycles (28 day Cycle)
  To determine the safety, tolerability and toxicity of CPX-351 in the maintenance setting for newly diagnosed AML in complete remission by analyzing the incidence of treatment emergent adverse events reported.
Overall Survival (Phase 1 and 2) | 1 year after end of treatment
  Determine the efficacy of CPX-351 as maintenance treatment in newly diagnosed AML patients who have achieved remission after induction treatment as measured by overall survival of subjects.
Event free survival (Phase 1 and 2) | 1 year after end of treatment
  Determine efficacy of CPX-351 as maintenance treatment in newly diagnosed AML patients who have achieved remission after induction treatment as measured by event free survival.
Relapse Free Survival (Phase 1 and 2) | 1 year after end of treatment
  Determine efficacy of CPX-351 as maintenance treatment in newly diagnosed AML patients who have achieved remission after induction treatment as measured by relapse free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Doucette, MD, Principal Investigator — Georgetown University
Locations (3):
- United States (3):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No